CLINICAL TRIAL: NCT01943019
Title: A Pilot Study to Assess the Efficacy of Linagliptin as an Adjunct in Schizophrenia Patients
Brief Title: Linagliptin in Schizophrenia Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inability to obtain patients
Sponsor: Monash University (Other)
Collaborators: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Shaun Lee Wen Huey, Dr, Monash University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Phamon 001
Record Dates: First submitted 2013-08-22; First posted 2013-09-16 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Linagliptin (Experimental): Linagliptin daily
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: Linagliptin

SUMMARY:
Approximately one third of patients with schizophrenia show a poor response to standard treatment with antipsychotic medications. This treatment resistant group of patients represents a major challenge in everyday psychiatry, and consumes a disproportionate amount of time from the clinicians, resulting in considerable costs to the society and government. Anecdotal evidence suggests that the enzyme dipeptidyl peptidase IV (DPPIV) may be altered in patients with schizophrenia, with a higher level DPPIV enzyme activity being noted. We postulate that this may play a role in the neuropathology of schizophrenia patients and by inhibiting the DPPIV enzyme activity with a DPPIV inhibitor such as linagliptin, we will be able to improve and even ameliorate the symptoms of schizophrenic patients. However, until now there have yet any studies on the potential of these inhibitors in schizophrenia patients. A pilot study is thus proposed to evaluate the potential of the DPPIV inhibitor, linagliptin as an adjunct in schizophrenia patients who are non-responsive to treatment, which will establish the feasibility of a larger trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and above
* Diagnosis of schizophrenia.
* Clinically stable antipsychotic regimen for the last 3 months
* A total score of 80 or greater at baseline on the Positive and Negative Syndrome Scale
* Competent and willing to provide written, informed consent

Exclusion Criteria:

* History of substance dependence within the past 2 months
* Existing relevant physical health problems: such as uncontrolled cardiovascular disease and impaired liver/ renal function
* History of diabetes
* History of hepatic or biliary diseases / biliary obstruction
* A serious suicide/homicide risk in the opinion of the investigator
* Known allergy to linagliptin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-08; Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
PANSS Score | 3 months

SECONDARY OUTCOMES:
Drug safety | 3 months
  No of adverse events recorded per patients

OTHER OUTCOMES:
DPP-4 enzyme levels | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Maniam Thambu, Principal Investigator — Pusat Perubatan UKM
Locations (1):
- Pusat Perubatan Universiti Kebangsaan Malaysia, Bandar Tun Razak, Kuala Lumpur, Malaysia